CLINICAL TRIAL: NCT04357496
Title: COVID-19 Epidemic Response Study: A National Observational Longitudinal Non-Interventional Protocol
Brief Title: COVID-19 Epidemic Response Study
Acronym: COVeR
Status: Withdrawn | Type: Observational
Why Stopped: study has never been started and was decided to be cancelled.
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: COVER-2020
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Fever; Pneumonia; Cough
Keywords: COVID-19
MeSH Terms: conditions — Fever; Pneumonia; Cough; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs and blood draws. Buccal swabs will be taken once per week within the first 4 weeks. Blood samples will be taken once a week for the first 6 weeks, and then once per month for the following 4.5 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with SARS-COV-2: Participants tested positive for SARS-COV-2 aged 60 years or older

SUMMARY:
A national, observational, longitudinal, non-interventional program aiming to identify prognostic parameters, to investigate the kinetics of the immune response, and to identify predictive biomarkers in SARS-CoV-2 infected patients.

DETAILED DESCRIPTION:
By 31st December 2019, 27 subjects with pneumonia of unknown aetiology were registered in Wuhan City, China. 7th of January the disease causative agent was identified and turned to be severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The WHO named the disease - coronavirus disease (COVID-19). On March 11, 2020, the World Health Organization (WHO) announced that COVID-19 should be characterized as a pandemic. At great economic cost, many countries have adopted unprecedented measures to curb the spread of the virus, such as large-scale use of isolation and quarantine, closing borders, imposing limits on public gatherings, and implementing nationwide lockdowns.

The most common symptoms of COVID-19 are fever, tiredness, and dry cough. Some patients may exhibit nasal congestion, runny nose, sore throat or diarrhea. These symptoms are usually mild and begin gradually. About 40% of the symptomatic patients recover from the disease without needing special treatment. Around 1 out of every 6 people infected with SARS-CoV-2 becomes seriously ill and develops difficulty breathing. Older people, and those with underlying medical problems like high chronic cardiovascular and respiratory disease or diabetes, are more likely to develop serious illness.

Monitoring patients with resolution of COVID-19 pneumonia is important in terms of when they should be released from isolation and discharged and to what extent this result is correlating with the clinical severity. If patients are still shedding viable coronavirus, they are likely to infect others. Therefore, quarantine for up to one month may be advisable. The optimal method for test of cure most likely will be two consecutive negative real-time RT-PCR tests. Furthermore, people who have cleared SARS-CoV-2 could have developed specific antibodies against the infectious agent in their blood plasma as a result of humoral immune response. This plasma is rich with specific antibodies and is called convalescent plasma (CP) or convalescent serum (CS). CP could treat and eradicate SARS-CoV-2 in infected individuals and could be used as therapy. This therapy concept was centuries old and was previously attempted during several outbreaks. Currently, there are few reports from China and South Korea showing that patients who received CP transfusion together with antiviral drugs and corticosteroids have recovered from the disease.

It is the aim of the COVeR study to enroll 400 patients with COVID-19 from nursing homes of the german state Mecklenburg-Vorpommern. Each patient will enter a follow-up phase of 6 months during which buccal swaps will be collected for judging the viral load, and blood samples for investigation of their immune response and identifying predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant/legal guardian
* Participant has been identified to be positive for SARS-C0V-2
* The participant is 60 years old or older

Exclusion Criteria:

* The informed consent is not obtained from the participant/legal guardian
* Participant has not been identified to be positive for SARS-C0V-2
* The participant is younger than 60 years of age

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with SARS-C0V-2
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Identification of prognostic parameters for SARS-CoV-2 infected participants. | 7 months
  Blood samples drawn from the infected participants will be analysed for prognostic parameters.

SECONDARY OUTCOMES:
Investigation of the kinetics of immune activation and antibody production against SARS-CoV-2 and correlation with clinical course | 7 months
  Systems from Abbott and Euroimmun will be used for IgG and IgM in SARS-CoV-2.

OTHER OUTCOMES:
Identification of predictive biomarker/s for clinical course in mildly and severely affected Covid-19 patients using genomic, proteomic, and transcriptomic approach. | 7 months
  Genomic, proteomic, and transcriptomic analyses will be performed on the blood samples drawn from Covid-19 infected participants over the course of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, Prof., Principal Investigator — CENTOGENE GmbH Rostock